CLINICAL TRIAL: NCT00123045
Title: Patient-Physician Partnership to Improve High Blood Pressure Adherence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 232; R01HL069403 (NIH); NCT00181324 (obsolete NCT alias)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: health education

SUMMARY:
To test the efficacy of a patient-centered, culturally tailored education and activation intervention designed to improve adherence to medication and life style recommendations among adults with uncontrolled hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension is a common, chronic condition that contributes substantially to cardiovascular morbidity and mortality and resource use. Despite the proven efficacy of pharmacologic therapy and lifestyle modification for treatment of hypertension and prevention of its complications, most adults with established hypertension are uncontrolled. Limited access to medical care and financial barriers to obtaining medications play an important role; however, even among patients who receive regular care, blood pressure control remains suboptimal. Patient non-adherence to recommended therapies and problems in physician management of patients with hypertension are critical contributors to poor quality of care and negative health outcomes of hypertension. Of particular concern is the disproportionately high prevalence and incidence of hypertension and its complications among African Americans and socioeconomically disadvantaged persons. Ethnic and social class disparities in patient adherence are frequently based on financial, logistical, environmental, and cultural barriers that, while not unique to ethnic minorities and the poor, have a greater impact on these populations. Patient and physician interventions were designed to address the specific needs of inner city ethnic minorities and persons living in poverty. The study used a patient-centered, culturally tailored, education and activation intervention with active follow-up delivered by a community health worker in the clinic. It also included a computerized, self-study communication skills training program delivered via an interactive CD-ROM, with tailored feedback to address physicians' individual communication skills needs.

DESIGN NARRATIVE:

The study used a patient-centered, culturally tailored, education and activation intervention with active follow-up delivered by a community health worker in the clinic. It also included a computerized, self-study communication skills training program delivered via an interactive CD-ROM, with tailored feedback to address physicians' individual communication skills needs. Fifty physicians and 500 of their patients who had uncontrolled hypertension were recruited into a randomized controlled trial with a 2X2 factorial design. The 50 physicians were randomized to receive either a 2-hour CD-ROM based communication skills training or no training. Within each randomized physician, 10 patient-subjects were randomized to either minimal intervention or patient activation (community health worker visit and follow-up calls, plus photo novels and other mailed educational literature). Assessments of primary care appointment keeping, medication possession, medication taking, health status, satisfaction, and numerous other variables were made at baseline, 3 months, and 12 months.

ELIGIBILITY:
Physicians - general internists and family physicians who see patients at least 20 hours per week at one of the participating study sites. Physicians are excluded if they intend to leave the practice within 12 months.

Patients - adults aged 18 years and older, with a diagnosis of hypertension (at least one claim with the ICD-9 code 401 in the preceding year), and able to provide contact information for themselves and at least one other person.

Patients who are too acutely ill, disoriented, or unresponsive to complete the baseline assessment and those with medical conditions that might limit their participation in the study (e.g., AIDS/HIV, schizophrenia, cancer (except skin), Alzheimer's or other form of dementia; end-stage renal disease, congestive heart failure, or active tuberculosis) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2001-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Patient adherence | 12 months
  self-report, Morisky measure

SECONDARY OUTCOMES:
Reduction in systolic blood pressure | 12 months
  change in systolic blood pressure from baseline to 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Cooper, MD, MPH, Principal Investigator — Johns Hopkins University